CLINICAL TRIAL: NCT00126503
Title: A Phase I/II Trial of BAY 43-9006 in Combination With Bevacizumab in Patients With Advanced Renal Cancer
Brief Title: Sorafenib Tosylate and Bevacizumab in Treating Patients With Advanced Kidney Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00066; NCI-2009-00066 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000434814; URO 470 (Other: Vanderbilt-Ingram Cancer Center); 6555 (Other: CTEP); U01CA099177 (NIH); P30CA068485 (NIH)
Record Dates: First submitted 2005-08-02; First posted 2005-08-04 (Estimated); Results first posted 2013-06-28 (Estimated); Last update posted 2015-01-15 (Estimated); Status verified 2014-09

CONDITIONS: Chromophobe Renal Cell Carcinoma; Clear Cell Renal Cell Carcinoma; Papillary Renal Cell Carcinoma; Recurrent Renal Cell Carcinoma; Sarcomatoid Renal Cell Carcinoma; Stage IV Renal Cell Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Bevacizumab; Sorafenib

ARMS (1):
- Treatment (bevacizumab and sorafenib tosylate) (Experimental): Phase I: Patients receive sorafenib PO twice daily on days 1-28 and bevacizumab IV over 30-90 minutes on days 1 and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Cohorts of 3-6 patients receive escalating doses of sorafenib and bevacizumab until the MTD is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity. An additional 6 patients are treated at the MTD.
  Phase II: Patients receive sorafenib PO once daily on days 1-28 and bevacizumab IV over 90 minutes on days 1 and 15 at the MTD in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Bevacizumab; Drug: Sorafenib Tosylate; Other: Pharmacological Study; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Biological: Bevacizumab — Given IV
  Other Names: Avastin; rhuMab-VEGF
Drug: Sorafenib Tosylate — Given PO
  Other Names: BAY 54-9085; Nexavar; SFN
Other: Pharmacological Study — Correlative studies
  Other Names: pharmacological studies
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase I/II trial studies the side effects and best dose of sorafenib tosylate and bevacizumab and to see how well they work in treating patients with advanced kidney cancer. Sorafenib tosylate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Monoclonal antibodies, such as bevacizumab, can block tumor growth by targeting certain cells. Bevacizumab and sorafenib tosylate may also stop the growth of tumor cells by blocking blood flow to the tumor. Giving sorafenib tosylate together with bevacizumab may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the tolerability and maximum tolerated dose of Sorafenib (sorafenib tosylate) when given orally in combination with Bevacizumab in patients with renal cell carcinoma (RCC). (Phase I) II. To estimate the objective response rate of advanced RCC receiving the combination therapy of Bevacizumab and Sorafenib. (Phase II) III. To estimate the progression-free survival of advanced renal cell carcinoma patients to Sorafenib (sorafenib tosylate) in combination with Bevacizumab. (Phase II)

SECONDARY OBJECTIVES:

I. To obtain fixed tissue in the form of paraffin blocks or unstained slides for evaluation of the following: von Hippel-Lindau tumor suppressor, E3 ubiquitin protein ligase (VHL) mutation status and phosphatase and tensin homolog (PTEN) mutation and/or expression status; VHL downstream proteins; Apoptosis and proliferation status; Microvascular density, and if able to process; kinase status- phosphorylation, inactive for mitogen-activated protein (MAP) kinase, v-akt murine thymoma viral oncogene homolog 1 (Akt) and kinase insert domain receptor (KDR) if feasible.

II. In situations where fresh tumor may be obtained prior to and/or following therapy (4 weeks)

1. Assess tumor baseline and changes in signal transduction - Raf-1 proto-oncogene, serine/threonine kinase (Raf), mitogen-activated protein kinase kinase (MEK), mitogen-activated protein kinase 1 (Erk), Erk phosphorylation, Akt phosphorylation status and Raf subcellular localization.
2. fms-related tyrosine kinase 1 (VEGFR1) (flk1) and kinase insert domain receptor (VEGFR2) (flt1/KDR) status and tissue vascular endothelial growth factor (VEGF).
3. Tumor cell apoptosis - marker of proliferation Ki-67 (Ki-67), transferase dUTP nick end labeling (TUNEL) staining, and expression levels of BH3 interacting domain death agonist (BH3) domain containing proteins.
4. Tumor blood vessel characteristics - microvessel density, fraction of immature tumor blood vessels, endothelial cell apoptosis.
5. Presence of VHL downstream proteins III. To relate changes in tumor perfusion and vascular permeability on serial arterial spin labeled (ASL) and dynamic contrast-enhanced (DCE)-magnetic resonance imaging (MRI) to clinical outcome and anti-tumor effects.

IV. Evaluate the pharmacokinetics of Sorafenib (alone and in combination) and bevacizumab in patients enrolled on the maximum tolerated dose (MTD) dose level of Sorafenib and bevacizumab representing the recommended phase II dose (RPTD) schedule (200mg once daily [QD] Sorafenib and 5 mg/kg intravenously [IV] Q 2 weeks of bevacizumab).

V. To determine the steady-state trough plasma concentration of Sorafenib and trough concentration of Bevacizumab and relate to toxicity and correlative endpoints.

VI. Serial analysis of circulating angiogenic cytokines (i.e. VEGF, angiopoeitin 2, basic fibroblast growth factor [bFGF], interleukin [IL]-8 etc) and association of findings with response, response duration and prediction of relapse.

OUTLINE: This phase I dose-escalation study followed by a phase II study.

PHASE I: Patients receive sorafenib tosylate orally (PO) twice daily on days 1-28 and bevacizumab intravenously (IV) over 30-90 minutes on days 1 and 15.

Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of sorafenib tosylate and bevacizumab until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity. An additional 6 patients are treated at the MTD.

PHASE II: Patients receive sorafenib tosylate PO once daily on days 1-28 and bevacizumab IV over 90 minutes on days 1 and 15 at the MTD in the absence of disease progression or unacceptable toxicity*.

[Note: *Patients may remain on protocol if only 1 of the drugs is stopped.]

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* PHASE I ELIGIBILITY CRITERIA
* Patients must have histological or cytological confirmation of renal cell carcinoma (clear cell, papillary, chromophobe, or sarcomatoid) not curable by standard approaches; tumor must be measurable by Response Evaluation Criteria In Solid Tumors (RECIST) criteria; nephrectomy prior to enrollment is not required
* Patients may not have had prior therapy with inhibitors of the mitogen-activated protein (MAP) kinase pathway or inhibitors of VEGF and/or its receptor signaling (VEGFR2)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Life expectancy of greater than 3 months
* Hemoglobin (Hgb) >= 9.0gm/dl (transfusions allowed prior to enrollment)
* White Blood Count >= 3,000/mm^3
* Absolute Granulocyte Count >= 1,200/mm^3
* Platelet Count >= 100,000/mm^3
* Serum creatinine =< 1.5 x upper limit of normal (ULN) or serum creatinine clearance (CrCl) >= 40ml/min (neither drug is cleared by the kidney)
* Total Bilirubin =< 1.5 x ULN
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 2.5 x ULN
* International normalized ratio (INR) =< 1.5 and activated partial thromboplastin time (aPTT) that is not greater than 1.3 times the ULN
* Urine Dipstick must show less then 1+ protein in urine or the patient will require 24 hour urine collection with total protein =< 1000 mg/24 hour
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document
* PHASE II ELIGIBILITY CRITERIA
* Patients enrolled on the phase II portion of the study will be required to have predominantly clear cell variant of renal cell carcinoma with less than 25% of any other histology (papillary or chromophobe or oncocytic); there must be histologic confirmation by treating center of either primary or metastatic lesion; patients must be willing to consent for obtaining tumor tissue blocks or unstained slides from prior biopsy or surgery; patients who participated in the Phase I part of the protocol will not be part of the accrual to the Phase II cohort
* Patients enrolled on the phase II portion of the study will be required to have measurable disseminated disease that is not curable by standard radiation therapy or surgery
* Previous nephrectomy is required with the following exceptions:

  * Primary tumor =< 5cm or
  * Extensive liver (> 30% of liver parenchymal) or multiple (> 5) bone metastases, or extensive extrarenal tumor or unresectable local/regional tumor extension making nephrectomy a clinically questionable and unreasonable procedure
* For the phase II study, patients will be allowed no more than one prior regimen containing a vaccine or cytokine based immunotherapy or chemotherapy for advanced disease
* Hgb >= 9.0gm/dl (transfusions allowed prior to enrollment)
* White Blood Count >= 3,000/mm^3 (phase II)
* Absolute Granulocyte Count >= 1,200/mm^3 (phase II)
* Platelet Count >= 100,000/mm^3 (phase II)
* Serum creatinine =< 1.5 x upper limit of normal (ULN) or serum creatinine clearance (CrCl) >= 40ml/min (neither drug is cleared by the kidney) (phase II)
* Total Bilirubin =< 1.5 x ULN (phase II)
* AST/ALT =< 2.5 x ULN
* INR =< 1.5
* Urine Dipstick must show less then 1+ protein in urine or the patient will require 24 hour urine collection with total protein =< 1000 mg/24 hour (phase II)
* No prior malignancy diagnosed within the past 3 years with the exception of non-melanoma skin cancers, melanoma in situ, carcinoma in situ of the cervix, ductal carcinoma in situ, and lobular carcinoma in situ; any prior malignancy must have a very likely cure rate (75% or greater)
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant while participating in this study, she should inform her treating physician immediately (phase II)
* Ability to understand and the willingness to sign a written informed consent document (phase II)

Exclusion Criteria:

* History or clinical evidence of central nervous system (CNS) disease, including primary brain tumor (participants with a history of meningioma are not excluded), seizures not controlled with standard medical therapy, any brain metastasis, or history of stroke within the prior 12 months; patients who have had a history of brain metastasis that have been resected or have had radiosurgery with no progression for more than 6 months are eligible if the Principle Investigator from the coordinating center is consulted and agrees
* Patients entered onto the phase II study may not have received more than one chemotherapy or immunotherapy regimen for Stage IV disease
* Patients may not have received chemotherapy or immunotherapy within 4 weeks of initiating treatment; patients will not have received a regimen containing a monoclonal antibody within 8 weeks of initiating treatment; toxicities from radiation must have resolved and a minimum of two weeks must pass prior to enrollment
* Patients may not have had prior anti-angiogenic therapy including, Sunitinib, VEGF Trap; prior Temsirilomus, Everolimus, Bevacizumab and Sorafenib will not be allowed; thalidomide or interferon (IFN) alpha are allowed either for adjuvant therapy or stage IV disease
* History of allergic reactions attributed to Chinese hamster ovary cell products, other recombinant human antibodies, or compounds of similar chemical or biologic composition to Sorafenib
* History of bleeding diathesis or coagulopathy
* A condition that impairs patient's ability to swallow pills will make patient ineligible
* No major surgical procedure, open biopsy or significant traumatic injury within 28 days prior to initiation of therapy on trial
* Anticipation of the need for major surgery during the course of the study
* Current or recent use (within 7 days of starting the study drugs) of full-dose of anticoagulants (except as required to maintain patency of preexisting, permanent indwelling IV catheters or for deep vein thrombosis [DVT] prophylaxis, for subjects receiving warfarin, INR should be =< 1.5) or thrombolytic agent
* Patients with uncontrolled hypertension; blood pressure must be =< 150/90 mmHg at the time of enrollment on a stable antihypertensive regimen
* Patients with clinically significant cardiovascular disease within 1 year prior to study entry

  * Uncontrolled hypertension
  * Myocardial infarction or unstable angina < 6 months prior to registration
  * New York heart association grade II or greater congestive heart failure, serious cardiac arrhythmia requiring medication (participants with controlled atrial arrhythmias are not excluded), unstable angina pectoris
  * Grade II or greater peripheral vascular disease
* Serious, non-healing wound, ulcer, or bone fracture
* Significant proteinuria (> 1000 mg protein/24 hours ) at baseline; subjects discovered to have >= 1+ proteinuria on dipstick should undergo a 24-hour urine collection, which should contain < 1000 mg protein/ 24 hours to be allowed participation in the study
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection requiring parental antibiotics, or psychiatric illness/social situations that would limit compliance with study requirements
* Patients taking cytochrome P450 enzyme-inducing antiepileptic drugs will be excluded (phenytoin, carbamazepine, Phenobarbital, rifampin, and St.John's Wort)
* Pregnant and lactating women are excluded from the study; breastfeeding should be discontinued while receiving therapy
* Human immunodeficiency virus (HIV)-positive patients receiving combination anti-retroviral therapy are excluded from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2005-05; Primary Completion 2011-10 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Sosman, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (5):
- United States (5):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Dana-Farber Harvard Cancer Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Phase I/II study was open 5/2005 through 12/2010.
Pre-assignment Details: 73 patients consented, 4 of whom were determined to be ineligible.
Groups:
- Phase I: Sorafenib will be taken orally twice daily beginning on day 1 and continued for 28 days which will be defined as a cycle. Bevacizumab will be administered once every 14 days (with up to a 3 day window before or after 14 days to allow for unforeseen scheduling problems) beginning on day 1.
- Phase II: Sorafenib will be taken orally once daily at 200 mg beginning on day -14 and continued for 28 days per cycle. There is no planned interruption. Bevacizumab 5mg/kg IV will be administered every 14 days (+/- 3 days) beginning on day 1.
Period: Overall Study
Arm/Group | Phase I | Phase II
Started | 48 | 21
Completed | 1 | 0
Not Completed | 47 | 21
Not completed — disease progression | 23 | 14
Not completed — Withdrawal by Subject | 0 | 1
Not completed — alternative therapy | 1 | 1
Not completed — other complicating disease | 4 | 1
Not completed — Death | 3 | 0
Not completed — Adverse Event | 13 | 3
Not completed — non-compliant | 1 | 0
Not completed — Physician Decision | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I | Phase II | Total
Number analyzed (Participants) | 48 | 21 | 69
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 35 | 19 | 54
  >=65 years | 13 | 2 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (1) | 58 (1) | 62 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 40 | 14 | 54
Region of Enrollment [Number; unit: participants]
  United States | 48 | 21 | 69

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of BAY 43-9006 (Sorafenib)in Combination With Bevacizumab (Phase I)
Description: The highest dose in milligrams (mg) of BAY 43-9006 (Sorafenib) in combination with Bevacizumab while maintaining tolerability. Cohorts of 3-6 patients received escalating doses of sorafenib and bevacizumab until the maximum tolerated dose (MTD) was achieved. The MTD is defined as the dose preceding that at which 2 or more of 6 patients experience dose-limiting toxicity during the initial cycle of therapy. DLTs include absolute neutrophil count (ANC) < 500/mm3 for > 7 days, ANC < 1000/mm3 with fever > 101 degrees Fahrenheit, platelet count < 50,000 mm3, and non-hematologic toxicity Common Toxicity Criteria (CTC) >= Grade 3.
Time Frame: at 28 days
Population: Patients enrolled to determine the safety of BAY 43-9006 (Sorafenib) in combination with Bevacizumab
Measure: Number; unit: mg
Groups:
- Phase I: Sorafenib will be taken orally twice daily beginning on day 1 and continued for 28 days which will be defined as a cycle. Bevacizumab will be administered once every 14 days (with up to a 3-day window before or after 14 days to allow for unforeseen scheduling problems) beginning on day 1.
Arm/Group | Phase I
Number analyzed (Participants) | 48
mg | 200

2. Secondary Outcome: Overall Survival
Description: Months from date on-study to expired or last date known alive
Time Frame: on-study to date of expired or last date known alive
Population: All treated patients available for determination of overall survival. No patients in the Phase I cohort moved to the Phase II cohort. No Phase II patients were in the Phase I cohort.
Measure: Median (Full Range); unit: months
Groups:
- Phase I: The highest dose in milligrams (mg) of BAY 43-9006 (Sorafenib) in combination with Bevacizumab while maintaining tolerability. The highest dose in milligrams/kilograms of body weight mg/kg of Bevacizumab in combination with BAY 43-9006 (Sorafenib) while maintaining tolerability.
Arm/Group | Phase I | Phase II
Number analyzed (Participants) | 48 | 21
months | 24 [1 to 73] | 25 [5 to 59]

3. Secondary Outcome: Progression-free Survival
Description: Duration of months of progression-free survival (PFS). Determined by months to progressive disease or to last date known alive without progressive disease.
Time Frame: on-study to date of progression or last date known alive without progression
Population: All patients who underwent treatment. No patients in the Phase I cohort moved to the Phase II cohort. No Phase II patients were in the Phase I cohort.
Measure: Median (Full Range); unit: months
Arm/Group | Phase I | Phase II
Number analyzed (Participants) | 48 | 21
months | 11 [1 to 56] | 15 [1 to 49]

4. Primary Outcome: Maximum Tolerated Dose of Bevacizumab in Combination With BAY 43-9006 (Sorafenib)(Phase I)
Description: The highest dose in milligrams (mg) of Bevacizumab in combination with BAY 43-9006 (Sorafenib) while maintaining tolerability. Cohorts of 3-6 patients received escalating doses of sorafenib and bevacizumab until the maximum tolerated dose (MTD) was achieved. The MTD is defined as the dose preceding that at which 2 or more of 6 patients experience dose-limiting toxicity during the initial cycle of therapy. DLTs include absolute neutrophil count (ANC) < 500/mm3 for > 7 days, ANC < 1000/mm3 with fever > 101 degrees Fahrenheit, platelet count < 50,000 mm3, and non-hematologic toxicity Common Toxicity Criteria (CTC) >= Grade 3.
Time Frame: at 28 days
Population: Patients enrolled to determine the safety of BAY 43-9006 (Sorafenib) in combination with Bevacizumab
Measure: Number; unit: mg/kg
Arm/Group | Phase I
Number analyzed (Participants) | 48
mg/kg | 5

5. Primary Outcome: Objective Response
Description: Objective response as determined by RECIST v. 1.0 (measurable lesions: complete response (CR) disappearance of target lesions, partial response (PR) > 30% decrease in the sum of the longest diameter (LD) of target lesions, progressive disease (PD) > 20% increase in the sum of the LD of target lesions or appearance of new lesions, stable disease (SD) neither sufficient decrease nor increase of the sum of smallest sum of the LD of target lesions)or last date known alive
Time Frame: Every 8 weeks to date of progression
Population: Patients available for measurement of response to treatment with regimen. 7 Phase I and 4 Phase II patients were not available for measurement of response, respectively: disease progression (5, 2), complicating disease (1, 0), death on-study (1, 0), toxicity (0, 1), and alternative treatment (0, 1). All were counted as clinical progression.
Measure: Number; unit: participants
Groups:
- Phase I: The highest dose in milligrams (mg) of BAY 43-9006 (Sorafenib) in combination with Bevacizumab while maintaining tolerability. The highest dose in milligrams/kilograms of body weight mg/kg of Bevacizumab in combination with BAY 43-9006 (Sorafenib) while maintaining tolerability. No Phase I patients moved to the Phase II cohort.
- Phase II: Sorafenib will be taken orally once daily at 200 mg beginning on day -14 and continued for 28 days per cycle. There is no planned interruption. Bevacizumab 5mg/kg IV will be administered every 14 days (+/- 3 days) beginning on day 1. No Phase II patients were in the Phase I cohort.
Arm/Group | Phase I | Phase II
Number analyzed (Participants) | 41 | 17
participants
  Complete Response | 0 [5 to 48] | 0
  Partial Response | 23 | 3
  Progressive Disease | 2 | 0
  Stable Disease | 16 | 14

ADVERSE EVENTS:
Arm/Group | Phase I | Phase II
Serious Adverse Events (participants affected / at risk) | 17/48 | 8/21
Other Adverse Events (participants affected / at risk) | 48/48 | 21/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I (N=48) | Phase II (N=21)
Edema-limb (General disorders) | 1 (1) | 0 (0)
Hemorrhage, pulmonary/upper respiratory-nose (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pain-chest wall (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
CNS cerebrovascular ischemia (Nervous system disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Musculoskeletal/soft tissue-Other (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Neuropathy - sensory (Nervous system disorders) | 1 (1) | 0 (0)
Pain-abdomen NOS (Gastrointestinal disorders) | 3 (3) | 1 (1)
Pain-joint (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Somnomolence/depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Cardiac ischemia/infarction (Cardiac disorders) | 3 (3) | 1 (1)
Hyperuricemia (Renal and urinary disorders) | 1 (1) | 0 (0)
Vascular-other (Vascular disorders) | 1 (1) | 0 (0)
Infection with unknown ANC-pancreas (Infections and infestations) | 1 (1) | 0 (0)
Infection with unknown ANC-lung (pneumonia) (Infections and infestations) | 1 (1) | 0 (0)
Death not associated with CTCAE term-Disease progression NOS (General disorders) | 2 (2) | 0 (0)
Fracture (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Supraventricular and nodal arrhythmia-atrial fibrillation (Cardiac disorders) | 1 (2) | 0 (0)
Thrombosis/thrombus/embolism (Vascular disorders) | 1 (1) | 0 (0)
Infection-Other (Infections and infestations) | 1 (1) | 0 (0)
Infection with Grade 1 or 2 neutrophils (ANC < 1.0 x 10e9/L)-skin (cellulitis) (Infections and infestations) | 2 (2) | 1 (1)
Hypertension (Vascular disorders) | 10 (10) | 1 (1)
Hyperbilirubinemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Wound complication, non-infectious (General disorders) | 0 (0) | 1 (1)
Obstruction, GI-gallbladder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cardiac General-other (Cardiac disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils-bone (osteomyelitis) (Infections and infestations) | 0 (0) | 1 (1)
Pain-back (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Perforation, GI-colon (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Supraventricular and nodal arrhythmia-atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC < 1.0 x 10e9/L) (General disorders) | 0 (0) | 1 (1)
stricture/stenosis (including anastomotic), GI-jejunum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oral mucositis (Gastrointestinal disorders) | 3 (3) | 0 (0)
palmar-plantar paresthesia (Skin and subcutaneous tissue disorders) | 10 (10) | 0 (0)
weight loss (Investigations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I (N=48) | Phase II (N=21)
allergic reaction/hypersensivity (Immune system disorders) | 0 (0) | 1 (1)
allergic rhinitis (Immune system disorders) | 18 (33) | 10 (10)
ALT/SGPT (serum glutamine pyruvic transminase) (Investigations) | 11 (28) | 4 (9)
Anorexia (Gastrointestinal disorders) | 28 (72) | 10 (11)
AST, SGOT (serum glutamine oxaloacetic transminase) (Investigations) | 11 (30) | 4 (9)
Bronchospasm-wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bruising (in absence of Grade 3/4 thromboctyopenia) (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (2)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
constipation (Gastrointestinal disorders) | 22 (38) | 8 (12)
Constitutional symptoms Other (General disorders) | 3 (5) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 19 (30) | 10 (13)
Creatinine (Metabolism and nutrition disorders) | 9 (24) | 2 (5)
Dehydration (Metabolism and nutrition disorders) | 3 (4) | 0 (0)
Dental-teeth (Gastrointestinal disorders) | 0 (0) | 2 (4)
Dermatology/Skin-Other (Skin and subcutaneous tissue disorders) | 14 (31) | 6 (16)
Diarrhea (Gastrointestinal disorders) | 33 (171) | 9 (29)
Distension/bloating, abdominal (Gastrointestinal disorders) | 4 (10) | 0 (0)
Dizziness (Nervous system disorders) | 11 (19) | 5 (5)
Dry eye syndrome (Eye disorders) | 4 (8) | 0 (0)
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 5 (8) | 4 (4)
Dry skin (Skin and subcutaneous tissue disorders) | 16 (26) | 7 (8)
Dysphagia (Gastrointestinal disorders) | 7 (12) | 3 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 10 (16) | 4 (6)
Edema head and neck (General disorders) | 3 (4) | 1 (1)
Edema limb (General disorders) | 7 (13) | 6 (6)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Extemity-lower (gait/walking) (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 38 (140) | 13 (37)
Fever (in the absence of neutropenia, with neutropenia defined as ANC < 1.0 x 10e9/L (General disorders) | 3 (3) | 2 (3)
fistula-GI anus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 18 (32) | 4 (5)
Flu-like syndrome (General disorders) | 3 (6) | 2 (2)
Flushing (Vascular disorders) | 4 (5) | 1 (1)
Gastrointestinal-Other (Gastrointestinal disorders) | 8 (14) | 1 (1)
hair loss-scalp or body (Skin and subcutaneous tissue disorders) | 5 (15) | 6 (6)
Heartburn, dyspepsia (Gastrointestinal disorders) | 21 (41) | 6 (9)
Hemoglobin (Infections and infestations) | 9 (30) | 3 (9)
Hemorrhage, GI-lower GI NOS (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hemorrhage, GI oral cavity (Gastrointestinal disorders) | 4 (6) | 4 (4)
Hemorrhage, GI rectum (Gastrointestinal disorders) | 4 (4) | 2 (2)
Hemorrhage, GU urinary (Renal and urinary disorders) | 0 (0) | 4 (4)
Hemorrhage, GU vaginal (Reproductive system and breast disorders) | 0 (0) | 1 (3)
Hemorrhage, pulmonary/upper respiratory-nose (Respiratory, thoracic and mediastinal disorders) | 15 (26) | 9 (13)
Hemorrhoids (Gastrointestinal disorders) | 9 (11) | 1 (1)
Hypercalcemia (Investigations) | 0 (0) | 1 (1)
Hypercholesterolemia (Metabolism and nutrition disorders) | 0 (0) | 1 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 11 (26) | 4 (40)
Hyperkalemia (Metabolism and nutrition disorders) | 5 (9) | 1 (2)
Hypertension (Vascular disorders) | 20 (54) | 15 (26)
Hypocalcemia (Metabolism and nutrition disorders) | 5 (8) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 3 (8) | 2 (5)
Hypokalemia (Metabolism and nutrition disorders) | 5 (8) | 4 (9)
Hyponatremia (Metabolism and nutrition disorders) | 11 (22) | 3 (24)
Infection-Other (Infections and infestations) | 0 (0) | 2 (3)
Infection with normal ANC or Grade 1 or 2 neutrophils-cellulitis (Infections and infestations) | 3 (3) | 0 (0)
Insomnia (Psychiatric disorders) | 11 (13) | 6 (6)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 0 (0) | 1 (4)
Memory impairment (Nervous system disorders) | 5 (6) | 1 (1)
Metabolic/laboratory-Other (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Mood alteration-agitation (Psychiatric disorders) | 0 (0) | 1 (1)
Mood alteration-anxiety (Psychiatric disorders) | 10 (12) | 2 (2)
Mood alteration-depression (Psychiatric disorders) | 10 (11) | 2 (2)
Mucositis/stomatitis-anus/rectum (functional/symptomatic) (Gastrointestinal disorders) | 3 (13) | 1 (1)
Mucositis/stomatitis-oral cavity (clinical exam) (Gastrointestinal disorders) | 23 (43) | 9 (10)
Muscle weakness, generalized or specific area-upper extremity/whole body/generalized (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Musculoskeletal/soft tissue-Other (Musculoskeletal and connective tissue disorders) | 5 (7) | 0 (0)
Nail changes (Skin and subcutaneous tissue disorders) | 5 (6) | 1 (1)
Nausea (Gastrointestinal disorders) | 25 (57) | 9 (23)
Neurology-Other (Nervous system disorders) | 0 (0) | 1 (2)
Neuropathy - sensory (Nervous system disorders) | 15 (42) | 5 (7)
Obesity (Metabolism and nutrition disorders) | 4 (8) | 3 (4)
Ocular/visual-Other (Eye disorders) | 0 (0) | 2 (2)
Otitis, middle ear (non-infectious) (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Pain-abdomen NOS (General disorders) | 17 (35) | 6 (11)
Pain-anus/rectum (General disorders) | 4 (5) | 0 (0)
Pain-back (General disorders) | 17 (30) | 8 (17)
Pain-bone (General disorders) | 4 (7) | 1 (2)
Pain-chest/thorax (General disorders) | 6 (6) | 4 (7)
Pain-dental/periodontal (General disorders) | 4 (9) | 0 (0)
Pain-Head/headache (Nervous system disorders) | 26 (53) | 13 (20)
Pain-joint (Musculoskeletal and connective tissue disorders) | 17 (35) | 6 (16)
Pain-oral cavity/gums (General disorders) | 8 (12) | 1 (1)
Pain-Other/NOS (General disorders) | 10 (14) | 4 (8)
Pain-pelvis (General disorders) | 0 (0) | 1 (2)
Pain-sinus (General disorders) | 4 (9) | 3 (3)
Pain-stomach (Gastrointestinal disorders) | 6 (10) | 0 (0)
Pain-throat, pharynx (Respiratory, thoracic and mediastinal disorders) | 10 (17) | 5 (11)
Platelets (Investigations) | 4 (18) | 1 (5)
Proteinuria (Renal and urinary disorders) | 11 (49) | 9 (56)
Pruritis (Skin and subcutaneous tissue disorders) | 10 (15) | 5 (7)
Pulmonary\upper respiratory-Other (Respiratory, thoracic and mediastinal disorders) | 8 (13) | 4 (6)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 18 (30) | 9 (15)
Rash acne/actiform (Skin and subcutaneous tissue disorders) | 13 (17) | 3 (3)
palmar/plantar paresthesia (Skin and subcutaneous tissue disorders) | 27 (195) | 17 (41)
Renal/Genitourinary-Other (Renal and urinary disorders) | 0 (0) | 2 (2)
Rigor, chills (General disorders) | 9 (13) | 6 (7)
Sweating/diphoresis (Skin and subcutaneous tissue disorders) | 5 (10) | 3 (4)
Syncope/fainting (Nervous system disorders) | 0 (0) | 1 (1)
Taste alteration (dysgeusia) (Nervous system disorders) | 14 (26) | 5 (6)
Thyroid function, low (hypothyroidism) (Endocrine disorders) | 0 (0) | 3 (3)
Uric acid, serum-high (hyperuricemia) (Renal and urinary disorders) | 0 (0) | 3 (3)
Urinary frequency/urgency (Renal and urinary disorders) | 5 (7) | 2 (4)
Vascular-other (Vascular disorders) | 0 (0) | 1 (1)
Vision-blurred vision (Eye disorders) | 8 (9) | 1 (1)
Vision-flashing lights/floaters (Eye disorders) | 0 (0) | 3 (3)
Voice changes/dysarthria (Respiratory, thoracic and mediastinal disorders) | 33 (58) | 14 (21)
Vomiting (Gastrointestinal disorders) | 16 (28) | 5 (9)
Weight loss (Investigations) | 26 (67) | 9 (19)
Alkaline phosphatase (Investigations) | 4 (6) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 4 (15)
Arthritis (non-septic) (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bicarbonate, serum-low (Investigations) | 0 (0) | 2 (6)
Hyperbilirubinemia (Investigations) | 3 (3) | 1 (2)
Burn (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Chelitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Endocrine other (Endocrine disorders) | 0 (0) | 1 (1)
Extrapyramidal/involuntary movement/restlessnes (Nervous system disorders) | 0 (0) | 1 (1)
Hemoglobinuria (Renal and urinary disorders) | 0 (0) | 2 (3)
Hiccoughs (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Infection with unknown ANC-cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Infection with unknown ANC-soft tissue (Infections and infestations) | 0 (0) | 2 (2)
Pain-breast (Reproductive system and breast disorders) | 3 (4) | 0 (0)
Pain-extremity. limb (Musculoskeletal and connective tissue disorders) | 16 (31) | 8 (20)
Pain-buttock (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain-muscle (Musculoskeletal and connective tissue disorders) | 10 (11) | 3 (3)
Pain-neck (General disorders) | 6 (6) | 3 (3)
Pain-skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Hypophosphatemia (Investigations) | 11 (54) | 5 (9)
Pain-scalp (Skin and subcutaneous tissue disorders) | 10 (12) | 1 (1)
Tumor pain (General disorders) | 3 (8) | 0 (0)
Watery eye (epiphora, tearing) (Eye disorders) | 3 (4) | 0 (0)
Weight gain (Metabolism and nutrition disorders) | 4 (5) | 0 (0)
Confusion (Psychiatric disorders) | 3 (3) | 0 (0)
Hypotension (Vascular disorders) | 3 (3) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils-external ear (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils-Eye NOS (Eye disorders) | 0 (0) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils-lung (pneumonia) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Infection with unknown ANC-stomach (Gastrointestinal disorders) | 0 (0) | 1 (1)
Infection with unknown ANC-wound (Infections and infestations) | 0 (0) | 1 (1)
Leak (including anastomatic)-GI-rectum (Gastrointestinal disorders) | 0 (0) | 1 (1)
Left ventricular systolic dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Occular surface disease (Eye disorders) | 0 (0) | 1 (1)
Partial prothrombin time (PTT) (Investigations) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Supraventricular and nodal arrhythmia-atrial tachycardia/paroxysmal atrial tachycardia (Cardiac disorders) | 0 (0) | 1 (2)
Telangiectasia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Triglyceride, serum-high (Investigations) | 0 (0) | 1 (2)
Infection with normal ANC or Grade 1 or 2 neutrophils-sinus (Infections and infestations) | 0 (0) | 2 (2)
Infection with normal ANC or Grade 1 or 2 neutrophils-upper airway NOS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pain-chest wall (General disorders) | 3 (3) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 3 (4)
Mucositis/stomatitis (functional/symptomatic)-Oral cavity (Infections and infestations) | 0 (0) | 7 (10)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
pneumonitis/pumonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Vessel injury-vein-extremity-limb (Vascular disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
To depict results of this Phases I/II study accurately, each phase was entered as an ARM to enable separation of the data by phase. Events reported in the Adverse Event and Serious Adverse Event sections include AEs and SAEs from Phase I and Phase II

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less